CLINICAL TRIAL: NCT04823845
Title: Plantar Wart Treatment Using Adapalene Gel
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study never received IRB approval.
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20.1175
Record Dates: First submitted 2021-03-05; First posted 2021-04-01 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Plantar Wart
Keywords: Wart; Adapalene
MeSH Terms: conditions — Warts

STUDY DESIGN:
Intervention Model Description: apply study treatment to single group of patients.
Masking Description: patient information will be kept secure and no individual identifiers will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Plantar Wart Treatment Using Adapalene Gel 0.1% (Experimental): patients treated for plantar warts with Adapalene 0.1% gel
  Interventions: Drug: Topical Adapalene Gel 0.1%

INTERVENTIONS:
Drug: Topical Adapalene Gel 0.1% — applying Adapalene Gel 0.1% to plantar warts topically

SUMMARY:
This study seeks to research the efficacy of Adapalene 0.1% gel as a cost effective and low risk treatment option for plantar warts of the foot. Patients that present/diagnosed in designated clinics with plantar warts will be offered the option of being treated with regular superficial debridements of the epidermis and twice a day application of adapalene gel 0.1% under occlusion. Patients will be followed until resolution.

DETAILED DESCRIPTION:
PROBLEM/BACKGROUND: Plantar warts are the result of a DNA virus called Human Papilloma Virus (HPV), specifically subtypes 1,2,4,27, and 57. Plantar warts are a common complaint among adults and children when standing, walking or running as they are on the weight-bearing surface of the foot. These cutaneous infections often occur when walking barefoot at public pools, sidewalks, bathhouses etc. and the epidermis becomes compromised. Surfaces carrying HPV is transmitted and infects the keratinocyte in the compromised skin and begins hyperplasia in the granular, prickle layers, and the dermal papillae. Histologically cell nuclei are eccentrically seen surrounded by koilocytes (halos). This manifests as a hyperkeratotic cutaneous lesion that is a dermal outpouching with break in normal skin lines, painful with lateral or direct pressure, and pin point bleeding. These lesions are often self limiting and resolve in time. However, patients often complain of pain and seek treatments.

Patients often try over the counter remedies with no avail, and then seek professional help for the issue. The standard of care for clinicians is often to use debridement with some form of keratolytic topical agent, such as: salicylic acid, canthridin is used; or cryotherapy, laser (pulse dye or CO2), bleomycin or candida injections are commonly used. Surgical excision is often utilized as well. These treatments are often invasive, painful, and require multiple sessions over a long period of time. Research has suggested the use of adapalene gel 0.1% as a less invasive and faster therapy for plantar warts. The purpose of this study is to test a United States population with Adapalene Gel 0.1% for plantar warts as a viable treatment option with the goals of being faster and less invasive.

OBJECTIVES: Test United States population in the treatment of plantar warts using adapalene gel 0.1%. Measure the amount of time until resolution of the plantar wart using this treatment. Document patient pain with this treatment method.

STUDY DESIGN: Clinician Interventional Prospective Study. Goal of minimum 50 patients will be studied from ages 5-90 years old of all health statuses, race, and genders. Pregnant women will be excluded due to very minimal, but medicine recommendations and guidelines. Patients presenting to outpatient clinics with plantar warts will be treated with a debridement with scalpel down to dermis followed by application of Adapalene 0.1% gel under occlusion. Patients will apply this twice a day under occlusion and return for repeat debridements every 2 weeks. Warts will be measured initially and before and after each debridement until resolution. Patient pain will be assessed each visit and documented.

SUBJECT RECRUITMENT: Patients will present to outpatient clinics, and if diagnosed with a plantar wart will be offered the standard of care treatment at that clinic or the Adapalene gel study treatment if they have not tried any other therapies for 2 weeks. Patients will have the option for the standard of care at the clinic or choose the treatment option of this study. Pregnant women will be excluded. Any patient having received another treatment therapy in the last 2 weeks will be excluded.

INFORMED CONSENT: Patients included in the study will be informed that this is not the standard of care, and that the standard of care is actually more invasive. This alternative treatment has been researched and has evidence to be safer, less invasive, and faster than the current standard of care. Patients will have the option to choose.

RESEARCH PROCEDURES: The research group will have their plantar warts photographed, pain assessed, measured, debrided down to the dermal layer using a sterile 15 scalpel, re-measured, apply adaplene 0.1% gel to area, cover with occlusive bandage. Patient will apply this adapelene gel 0.1% twice a day daily and keep covered at all times.

STATISTICAL ANALYSIS: Descriptive and inferential statistics will be calculated on 50 patients recruited into the study who had plantar warts. Measures taken will be the age and sex of patients, duration of warts in months, size of warts, time taken to remove the warts by using Adapalene gel 0.1% under occlusion, and side effects of usage such as irritation, erethyma, and scar tissue. Statistics will include frequency and percentages, and means ± standard deviations where appropriate. Confidence intervals (95 CIs) will be calculated around the time taken to remove the warts. A sample size and power analysis showed that if the mean time to remove the warts using Adapalene gel was 37 days with a standard deviation of 19, a sample size of 50 would allow us to obtain 95% CIs of 31.6, 42.4 days." RESEARCH MATERIALS: Patient's age, gender, race, BMI will be recorded in the EMR as well as wart size, photo, and pain level each visit.

ELIGIBILITY:
Inclusion Criteria:

* patients must be diagnosed with plantar warts

Exclusion Criteria:

* pregnant women
* previous wart treatment within the last 2 weeks

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
Time Until Plantar Wart Resolution | 30-60 days
  days

IPD SHARING:
Plan to Share IPD: No
IPD will only be obtained/used by the researchers and no individual patient identifiers will be used.

REFERENCES:
- [Background] Gupta R, Gupta S. Topical adapalene in the treatment of plantar warts; randomized comparative open trial in comparison with cryo-therapy. Indian J Dermatol. 2015 Jan-Feb;60(1):102. doi: 10.4103/0019-5154.147835. PMID 25657417
- [Background] Gupta R. Plantar warts treated with topical adapalene. Indian J Dermatol. 2011 Sep-Oct;56(5):513-4. doi: 10.4103/0019-5154.87135. PMID 22121266
- [Background] Vlahovic TC, Khan MT. The Human Papillomavirus and Its Role in Plantar Warts: A Comprehensive Review of Diagnosis and Management. Clin Podiatr Med Surg. 2016 Jul;33(3):337-53. doi: 10.1016/j.cpm.2016.02.003. Epub 2016 Mar 29. PMID 27215155